CLINICAL TRIAL: NCT02101216
Title: A Randomized, Open-Label, Single-Dose, 2 Period Crossover Pharmacokinetic and Bioequivalence Study, With a Lead-In Dose Period, Evaluating Oral Abacavir Acetate (Prurisol™) and Oral Abacavir Sulfate (Ziagen®) in Healthy Volunteers
Brief Title: Bioequivalence and Pharmacokinetic Study of Prurisol™ and Abacavir Sulfate in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cellceutix Corporation (Industry)
Responsible Party: Sponsor
Organization: Innovation Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CTIX-14-03
Record Dates: First submitted 2014-03-24; First posted 2014-04-02 (Estimated); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Psoriasis
Keywords: bioequivalence; pharmacokinetics; psoriasis
MeSH Terms: conditions — Psoriasis | interventions — abacavir hydroxyacetate; abacavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Pharmacokinetics of low dose Prurisol (Experimental): Pharmacokinetics of single dose of Prurisol™ 50 mg (1 tablets) to 6 subjects
  Interventions: Drug: Prurisol
- Pharmacokinetics medium dose Prurisol (Experimental): Pharmacokinetics of single dose of Prurisol™ 100 mg (2 tablets) to 6 subjects
  Interventions: Drug: Prurisol
- Pharmacokinetics of high dose Prurisol (Experimental): Pharmacokinetics of single dose of Prurisol™ 200 mg (4 tablets) to 6 subjects
  Interventions: Drug: Prurisol
- Bioequivalence of Prurisol (350 mg) (Experimental): Single dose of Prurisol™ 350 mg (7 x 50 mg tablets)
  Interventions: Drug: Prurisol
- Bioequivalence of Ziagen (300 mg) (Active Comparator): Single dose of Ziagen 300 mg (1 x 300mg tablet)
  Interventions: Drug: Ziagen

INTERVENTIONS:
Drug: Prurisol — Experimental Drug
  Other Names: abacavir acetate
  Arms: Bioequivalence of Prurisol (350 mg); Pharmacokinetics medium dose Prurisol; Pharmacokinetics of high dose Prurisol; Pharmacokinetics of low dose Prurisol
Drug: Ziagen — Active comparator
  Other Names: abacavir sulfate
  Arms: Bioequivalence of Ziagen (300 mg)

SUMMARY:
Cellceutix Corporation has created a new chemical entity for the treatment of psoriasis, termed Prurisol™, which is an ester of abacavir. This first-in-human study of Prurisol (abacavir acetate) is being performed to evaluate the pharmacokinetics, safety and tolerance of a single oral doses of Prurisol administered to healthy volunteers and the bioequivalence to abacavir sulfate (Ziagen). This study will be followed by a 505(b)(2) Phase 2 trial in patients with moderate to severe plaque psoriasis.

DETAILED DESCRIPTION:
Prurisol™, abacavir acetate, is an ester of abacavir. Prurisol is believed to act as an immune response modifier in certain conditions, including psoriasis. Abacavir is a synthetic nucleoside analogue. Ziagen, abacavir sulfate, was developed and marketed as a treatment for HIV-1 infection for over a decade. Ziagen inhibits viral DNA synthesis. Consequently, Prurisol is under consideration as a possible new therapy for moderate to severe plaque psoriasis. The nonclinical efficacy of Prurisol has been demonstrated in the human psoriatic skin xenograft model in irradiated severe combined immune deficient mice. Histologic as well as visual observations confirmed a treatment benefit of Prurisol in this animal model. Interleukin-20 (IL-20) is a recently discovered cytokine displaying increased levels in psoriatic lesions, and levels of IL-20 have been shown to decrease with anti-psoriasis treatment and correlate with clinical improvement. IL-20 has been suggested as a specific target in psoriasis treatment. In comparison to vehicle-treated animals, the mice transplanted with human psoriatic tissue and treated with Prurisol had significant reductions in plasma IL-20 levels which were greater than those seen with methotrexate treatment. The expression of PRINS (psoriasis susceptibility-related RNA gene induced by stress) was significantly lower with twice daily Prurisol treatment compared to control.

This study is designed as an open-label, randomized, 2-period, 2-treatment, 2-sequence, single-dose intensive pharmacokinetic (PK) study conducted in healthy volunteers. In addition, a lead-in dosing period will allow the evaluation of the PK of abacavir from 3 escalating single doses of Prurisol (50mg, 100mg, 200mg). Completion of each dosing cohort will be followed by a 24-hour safety evaluation period before moving to a higher dose. Adverse Events, vital signs, physical examination, and safety laboratory tests (clinical chemistry and hematology) from each dosed cohort will be reviewed prior to any dose escalation for next cohort.

For each subject completing the first part, there will be a 5 to 21 day washout period before the next dose of study drug. Subjects will be randomly assigned to receive either a single dose of 350mg Prurisol or 300mg of Ziagen in the second dosing period. After a 5 to 21 day washout period, subjects will receive the alternate treatment in the third dosing period.

Blood samples for PK analysis will be obtained over a 24 hour period for each dose. Safety and tolerability will be assessed by ascertainment of adverse events, results of clinical laboratory testing and physical examination.

ELIGIBILITY:
Inclusion Criteria:

Individuals who meet ALL of the following criteria are eligible for participation in this study:

* Provided written informed consent
* Male or female adult aged 18-65 years old (inclusive). At least 20% of enrolled subjects will be aged 55-65 years, inclusive. Effort will be made to enroll equivalent numbers of males and females
* BMI of 19-32 kg/m2
* Identified as a non-smoker at the Consent/Screening Visit. A urine cotinine test will be performed at screening and during each clinic check-in before for each of the three Treatment Visits
* Willing and able to comply with all aspects of the study protocol including avoiding use of certain concomitant medications and attending the required clinic visits

Exclusion Criteria:

Subjects are not eligible for participation in the study if any of the following criteria are met:

* Females of childbearing potential not using reliable contraception, (e.g., abstinence, double barrier method, oral/implantable/transdermal contraception. Depo-provera, intrauterine device)
* Female who is pregnant, lactating, has a positive serum pregnancy test drawn at the Consent/Screening Visit, or has a positive urine pregnancy test at check-in performed prior to any of the 3 Treatment Days
* Presence of any uncontrolled (in the Investigator's medical opinion) systemic disease, including, but not limited to renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, or psychiatric disease
* History of any immune disorder, or disease/condition potentially affecting the immune system
* Regular use of oral or parenteral corticosteroids (inhaled corticosteroids for stable asthma or chronic obstructive pulmonary disease are permitted)
* ECG obtained at Consent/Screening Visit which shows medically significant abnormalities (e.g. bundle branch block, frequent premature ventricular contractions, corrected QT interval (QTc) prolongation >450 msec for males and >470 msec for females)
* Presence of a condition that makes it unlikely that the requirements of the protocol will be completed
* Urine screening test(s) positive for evidence of amphetamines, barbiturates, benzodiazepines, cocaine, methamphetamine, opiates, phencyclidine, marijuana
* Positive urine cotinine test
* Positive breath alcohol test
* History of hypersensitivity to any formulation of abacavir
* Previous treatment with any abacavir-containing product
* Current participation or participation in a drug/device or biologic investigational research study within 30 days prior to the Treatment A Visit
* An elective surgical or medical procedure is planned or scheduled to be performed during the period of the study
* Past surgical history of any degree of gastric resection or gastric banding
* History of a clinically diagnosed upper respiratory tract infection or any acute illness requiring antibiotic therapy within 14 days prior to the Treatment A Visit
* Systolic blood pressure >150 mmHg or diastolic blood pressure >90 mmHg or heart rate <45 bpm in a subject under the age of 40 years and heart rate <50 bpm in a subject aged ≥40 years or >100 bpm (any subject age) on repeat determinations at the Consent/Screening Visit or at check-in on the day prior to each of the 3 Treatment Days and at pre-dose if drug administered on different day than check-in
* Clinical laboratory results at the Consent/Screening Visit that show any one or more of the following:

  * Hemoglobin <11 Gm/dL, Hematocrit<30%
  * Total white blood cell count <3000cells/mm3
  * Absolute neutrophil count <1500cells/mm3
  * Platelet count <100,000/mm3
  * alanine aminotransferase or aspartate aminotransferase >1.5 x Upper Limit of Normal (ULN)
  * Serum amylase above ULN
  * Serum creatinine >1.5 x ULN
  * Positive serum human chorionic gonadotropin
  * Positive serologic test for HBsAg, HIV, hepatitis C virus
  * Positive test for HLA-B*5701 allele by certified laboratory
  * Urinalysis showing medically significant abnormality

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-03; Primary Completion 2014-07 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of abacavir derived from Prurisol and Ziagen | 24 hours after second and third dose of study drug or reference drug
  Part B of the study will determine the average bioequivalence of abacavir derived from Prurisol (abacavir acetate) 350mg compared with abacavir derived from the commercially available tablet formulation of Ziagen (abacavir sulfate) 300mg.
  After completion of Part A, subjects will be randomly assigned to cross-over treatment sequence Prurisol then Ziagen, or Ziagen then Prurisol. Five to 21 days later, each subject will receive the alternate study drug. Evaluable subjects in the PK population will be those who received both alternate treatments and for whom an adequate number of post-dose PK sample results are available.
Peak plasma concentration (Cmax) of abacavir derived from Prurisol and Ziagen | 24 hours after second and third dose of study drug or reference drug
  Part B of the study will determine the average bioequivalence of abacavir derived from Prurisol (abacavir acetate) 350mg compared with abacavir derived from the commercially available tablet formulation of Ziagen (abacavir sulfate) 300mg.
  After completion of Part A, subjects will be randomly assigned to cross-over treatment sequence Prurisol then Ziagen, or Ziagen then Prurisol. Five to 21 days later, each subject will receive the alternate study drug. Evaluable subjects in the PK population will be those who received both alternate treatments and for whom an adequate number of post-dose PK sample results are available.
Time to Cmax (Tmax) of abacavir derived from Prurisol and Ziagen | 24 hours after second and third dose of study drug or reference drug
  Part B of the study will determine the average bioequivalence of abacavir derived from Prurisol (abacavir acetate) 350mg compared with abacavir derived from the commercially available tablet formulation of Ziagen (abacavir sulfate) 300mg.
  After completion of Part A, subjects will be randomly assigned to cross-over treatment sequence Prurisol then Ziagen, or Ziagen then Prurisol. Five to 21 days later, each subject will receive the alternate study drug. Evaluable subjects in the PK population will be those who received both alternate treatments and for whom an adequate number of post-dose PK sample results are available.

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of abacavir derived from Prurisol | 0 to 24 hours after the first dose of study drug
  Pharmacokinetic parameters (AUC, Cmax, Tmax, t1/2) of abacavir derived from Prurisol will be determined in Part A of this study. Three cohorts, each comprising 6 subjects, will be administered escalating single doses of Prurisol.
  Part A consists of single doses of open-label Prurisol at doses of 50mg (1 tablet), 100mg (2 tablets) and 200 mg (4 tablets) administered to approximately equal numbers of male and female subjects. These treatments will be administered in 3 sequential cohorts with at least a 24 hour interval (safety period) between subjects in each of the 3 cohorts.
  Plasma concentrations of abacavir will be assayed by a validated liquid chromatography-mass spectrometry (LC/MS/MS) method and PK parameters will be calculated.
Peak plasma concentration (Cmax) of abacavir derived from Prurisol | 0 to 24 hours after the first dose of study drug
  Pharmacokinetic parameters (AUC, Cmax, Tmax, t1/2) of abacavir derived from Prurisol will be determined in Part A of this study. Three cohorts, each comprising 6 subjects, will be administered escalating single doses of Prurisol.
  Part A consists of single doses of open-label Prurisol at doses of 50mg (1 tablet), 100mg (2 tablets) and 200 mg (4 tablets) administered to approximately equal numbers of male and female subjects. These treatments will be administered in 3 sequential cohorts with at least a 24 hour interval (safety period) between subjects in each of the 3 cohorts.
  Plasma concentrations of abacavir will be assayed by a validated liquid chromatography-mass spectrometry (LC/MS/MS) method and PK parameters will be calculated.
Time to Cmax (Tmax) of abacavir derived from Prurisol | 0 to 24 hours after the first dose of study drug
  Pharmacokinetic parameters (AUC, Cmax, Tmax, t1/2) of abacavir derived from Prurisol will be determined in Part A of this study. Three cohorts, each comprising 6 subjects, will be administered escalating single doses of Prurisol.
  Part A consists of single doses of open-label Prurisol at doses of 50mg (1 tablet), 100mg (2 tablets) and 200 mg (4 tablets) administered to approximately equal numbers of male and female subjects. These treatments will be administered in 3 sequential cohorts with at least a 24 hour interval (safety period) between subjects in each of the 3 cohorts.
  Plasma concentrations of abacavir will be assayed by a validated liquid chromatography-mass spectrometry (LC/MS/MS) method and PK parameters will be calculated.
Elimination half-life (t1/2) of abacavir derived from Prurisol | 0 to 24 hours after the first dose of study drug
  Pharmacokinetic parameters (AUC, Cmax, Tmax, t1/2) of abacavir derived from Prurisol will be determined in Part A of this study. Three cohorts, each comprising 6 subjects, will be administered escalating single doses of Prurisol.
  Part A consists of single doses of open-label Prurisol at doses of 50mg (1 tablet), 100mg (2 tablets) and 200 mg (4 tablets) administered to approximately equal numbers of male and female subjects. These treatments will be administered in 3 sequential cohorts with at least a 24 hour interval (safety period) between subjects in each of the 3 cohorts.
  Plasma concentrations of abacavir will be assayed by a validated liquid chromatography-mass spectrometry (LC/MS/MS) method and PK parameters will be calculated.
Number of participants with adverse events | Day 1, Day 2, Day 3
  To evaluate the safety and tolerability of Prurisol in healthy volunteers, completion of each dosing cohort will be followed by a 24-hour safety evaluation period before moving to a higher dose. Adverse events from each dosed cohort will be reviewed prior to any dose escalation for next cohort.
  For each subject completing their first treatment, there will be a 5 to 21 day washout period before being given the next dose of study drug. Subjects completing their first treatment will be randomly assigned to receive either Prurisol or Ziagen in the second dosing period. After a 5-21 day washout period, subjects will receive the alternate treatment (Ziagen or Prurisol) in the third dosing period.
  The sequential dosing specified will allow for observation of any possible adverse effects of Prurisol at the respective doses.
Number of participants with vital sign changes | Day 1, Day 2, Day 3
  To evaluate the safety and tolerability of Prurisol in healthy volunteers, completion of each dosing cohort will be followed by a 24-hour safety evaluation period before moving to a higher dose. Vital signs from each dosed cohort will be reviewed prior to any dose escalation for next cohort.
  For each subject completing their first treatment, there will be a 5 to 21 day washout period before being given the next dose of study drug. Subjects completing their first treatment will be randomly assigned to receive either Prurisol or Ziagen in the second dosing period. After a 5-21 day washout period, subjects will receive the alternate treatment (Ziagen or Prurisol) in the third dosing period.
  The sequential dosing specified will allow for observation of any possible adverse effects of Prurisol at the respective doses.
Number of participants with changes in standard laboratory tests | Day 1, Day 2, Day 3
  To evaluate the safety and tolerability of Prurisol in healthy volunteers, completion of each dosing cohort will be followed by a 24-hour safety evaluation period before moving to a higher dose. Laboratory tests (standard hematology and clinical chemistry panels) from each dosed cohort will be reviewed prior to any dose escalation for next cohort.
  For each subject completing their first treatment, there will be a 5 to 21 day washout period before being given the next dose of study drug. Subjects completing their first treatment will be randomly assigned to receive either Prurisol or Ziagen in the second dosing period. After a 5-21 day washout period, subjects will receive the alternate treatment (Ziagen or Prurisol) in the third dosing period.
  The sequential dosing specified will allow for observation of any possible adverse effects of Prurisol at the respective doses.

CONTACTS AND LOCATIONS:
Overall Officials: Krishna Menon, Study Director — Cellceutix Corporation
Locations (1):
- Phase One Solutions Inc., Miami Gardens, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Foster RH, Faulds D. Abacavir. Drugs. 1998 May;55(5):729-36; discussion 737-8. doi: 10.2165/00003495-199855050-00018. PMID 9585869
- [Background] Galadari I, Rigel E, Lebwohl M. The cost of psoriasis treatment. J Eur Acad Dermatol Venereol. 2001 Jul;15(4):290-1. No abstract available. PMID 11730031
- [Background] Hetherington S, McGuirk S, Powell G, Cutrell A, Naderer O, Spreen B, Lafon S, Pearce G, Steel H. Hypersensitivity reactions during therapy with the nucleoside reverse transcriptase inhibitor abacavir. Clin Ther. 2001 Oct;23(10):1603-14. doi: 10.1016/s0149-2918(01)80132-6. PMID 11726000
- [Background] Imamichi T. Action of anti-HIV drugs and resistance: reverse transcriptase inhibitors and protease inhibitors. Curr Pharm Des. 2004;10(32):4039-53. doi: 10.2174/1381612043382440. PMID 15579086
- [Background] Sonkoly E, Bata-Csorgo Z, Pivarcsi A, Polyanka H, Kenderessy-Szabo A, Molnar G, Szentpali K, Bari L, Megyeri K, Mandi Y, Dobozy A, Kemeny L, Szell M. Identification and characterization of a novel, psoriasis susceptibility-related noncoding RNA gene, PRINS. J Biol Chem. 2005 Jun 24;280(25):24159-67. doi: 10.1074/jbc.M501704200. Epub 2005 Apr 26. PMID 15855153
- [Background] Tzu J, Kerdel F. From conventional to cutting edge: the new era of biologics in treatment of psoriasis. Dermatol Ther. 2008 Mar-Apr;21(2):131-41. doi: 10.1111/j.1529-8019.2008.00180.x. PMID 18394087
- See also: Ziagen® Highlights of Prescribing Information — http://www.accessdata.fda.gov/drugsatfda_docs/label/2008/020977s019,020978s022lbl.pdf
- See also: Ziagen® NDA # 020977 (December 1998), — http://www.accessdata.fda.gov/scripts/cder/drugsatfda/index.cfm?fuseaction=Search.DrugDetails.
- See also: CDER FDA Guidance for Industry (January 2001). Statistical Approaches to Establishing Bioequivalence — http://www.fda.gov/downloads/Drugs/Guidances/ucm070244.pdf